CLINICAL TRIAL: NCT00851318
Title: A Multicenter, Open-label, Long-term Safety Study of CDP870 to Evaluate the Safety and Efficacy of CDP870 Administered in Combination With Methotrexate (MTX) Over the Long Term in Patients With Active Rheumatoid Arthritis Transferred From the Efficacy Confirmatory Study (Study 275-08-001)
Brief Title: Long-term Treatment Study of Certolizumab Pegol (CDP870) as Add-on Medication to Methotrexate in Japanese Rheumatoid Arthritis (RA) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDP870-275-08-002; JapicCTI-090700
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Certolizumab Pegol; Cimzia
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Certolizumab pegol 200 mg (Experimental): Participants received 200 mg certolizumab pegol by subcutaneous injection once every 2 weeks in combination with methotrexate for up to 52 weeks or until approval of certolizumab pegol for rheumatoid arthritis in Japan.
  Interventions: Drug: Certolizumab pegol; Drug: Methotrexate
- Certolizumab pegol 400 mg (Experimental): Participants received 400 mg certolizumab pegol by subcutaneous injection once every 4 weeks in combination with methotrexate for up to 52 weeks or until approval of certolizumab pegol for rheumatoid arthritis in Japan.
  Interventions: Drug: Certolizumab pegol; Drug: Methotrexate

INTERVENTIONS:
Drug: Certolizumab pegol — Subcutaneous (SC) injection
  Other Names: CDP870; Cimzia
Drug: Methotrexate — Methotrexate dose between 6 to 8 mg/week.

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy of certolizumab pegol as add-on medication to methotrexate over the long term in Japanese RA patients transferred from Study 275-08-001 (NCT00791999), and to evaluate the effects of different dosing regimens on the safety and efficacy of certolizumab pegol in American College of Rheumatology 20% (ACR20) responders who completed Study 275-08-001.

DETAILED DESCRIPTION:
This study was initiated by Otsuka Pharmaceutical Co., Ltd and transferred to Astellas on 12/04/2012.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who participated in Study 275-08-001 and meet all of the criteria described below.

  * Patients who did not reach ACR20, and prematurely discontinued Study 275-08-001 at Week 16 or completed Study 275-08-001 by Week 24.
  * Patients who are able to receive treatment with MTX, by Week 52.

Exclusion Criteria:

* Patients who experienced an important protocol deviation as mentioned below during Study 275-08-001.
* Patients who received live or attenuated vaccines during Study 275-08-001(Except for influenza or pneumococcal vaccines).
* Patients who were found to have tuberculosis on a chest X-ray during Study 275-08-001.
* Patients who required treatment for the same infection at two or more different times during Study 275-08-001
* Women who are pregnant, are lactating, of childbearing potential and wish to conceive during the study and post-study 3 months.
* Patients whom the investigator has decided to be inappropriate for participation in the study

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2009-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with rheumatoid arthritis (RA) who participated in Study 275-08-001 (NCT00791999) were eligible for this study.
Pre-assignment Details: Participants were assigned to treatment groups based on whether they discontinued study 275-08-001 at Week 16 or completed Week 24 and based on American College of Rheumatology 20% (ACR20) response at Week 24.
Groups:
- Discontinued Non-responders 200 mg: Participants who were ACR20 non-responders and discontinued study 275-08-001 at Week 16 received 200 mg certolizumab pegol by subcutaneous injection once every 2 weeks in combination with methotrexate for up to 52 weeks or until approval of certolizumab pegol for rheumatoid arthritis in Japan.
- Completed Non-responders 200 mg: Participants who were ACR20 non-responders and completed study 275-08-001 at Week 24 received 200 mg certolizumab pegol by subcutaneous injection once every 2 weeks in combination with methotrexate for up to 52 weeks or until approval of certolizumab pegol for rheumatoid arthritis in Japan.
- Completed Responders 200 mg: Participants who were ACR20 responders and completed study 275-08-001 at Week 24 received 200 mg certolizumab pegol by subcutaneous injection once every 2 weeks in combination with methotrexate for up to 52 weeks or until approval of certolizumab pegol for rheumatoid arthritis in Japan.
- Completed Responders 400 mg: Participants who were ACR20 responders and completed study 275-08-001 at Week 24 received 400 mg certolizumab pegol by subcutaneous injection once every 4 weeks in combination with methotrexate for up to 52 weeks or until approval of certolizumab pegol for rheumatoid arthritis in Japan.
Period: Overall Study
Arm/Group | Discontinued Non-responders 200 mg | Completed Non-responders 200 mg | Completed Responders 200 mg | Completed Responders 400 mg
Started | 81 | 19 | 93 | 92
Completed Week 24 | 69 | 17 | 90 | 87
Completed Week 52 | 64 | 16 | 87 | 85
Completed | 51 | 14 | 72 | 73
Not Completed | 30 | 5 | 21 | 19
Not completed — Withdrawal by Subject | 7 | 1 | 5 | 3
Not completed — Adverse Event | 13 | 2 | 9 | 12
Not completed — Pregnancy | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 8 | 2 | 4 | 2
Not completed — Non-compliance with Study Procedures | 2 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Discontinued Non-responders 200 mg: Participants who were non-responders and discontinued study 275-08-001 at Week 16 received 200 mg certolizumab pegol by subcutaneous injection once every 2 weeks in combination with methotrexate for up to 52 weeks or until approval of certolizumab pegol for rheumatoid arthritis in Japan.
- Completed Non-responders 200 mg: Participants who were non-responders and completed study 275-08-001 at Week 24 received 200 mg certolizumab pegol by subcutaneous injection once every 2 weeks in combination with methotrexate for up to 52 weeks or until approval of certolizumab pegol for rheumatoid arthritis in Japan.
- Completed Responders 200 mg: Participants who were responders and completed study 275-08-001 at Week 24 received 200 mg certolizumab pegol by subcutaneous injection once every 2 weeks in combination with methotrexate for up to 52 weeks or until approval of certolizumab pegol for rheumatoid arthritis in Japan.
- Completed Responders 400 mg: Participants who were responders and completed study 275-08-001 at Week 24 received 400 mg certolizumab pegol by subcutaneous injection once every 4 weeks in combination with methotrexate for up to 52 weeks or until approval of certolizumab pegol for rheumatoid arthritis in Japan.
- Total: Total of all reporting groups
Arm/Group | Discontinued Non-responders 200 mg | Completed Non-responders 200 mg | Completed Responders 200 mg | Completed Responders 400 mg | Total
Number analyzed (Participants) | 81 | 19 | 93 | 92 | 285
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (10.7) | 51.3 (13.7) | 52.9 (11.0) | 54.1 (11.0) | 52.8 (11.1)
Age, Customized [Number; unit: participants]
  < 65 years | 72 | 16 | 81 | 76 | 245
  ≧ 65 years | 9 | 3 | 12 | 16 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 16 | 76 | 77 | 236
  Male | 14 | 3 | 17 | 15 | 49
Region of Enrollment [Number; unit: participants]
  Japan | 81 | 19 | 93 | 92 | 285
Body Weight [Mean (Standard Deviation); unit: kg] | 56.30 (12.00) | 54.27 (9.57) | 55.81 (11.34) | 54.92 (9.47) | 55.56 (10.83)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered study drug which did not necessarily have a causal relationship with the treatment. In this study, events that occurred between the time of informed consent and the start of study medication were included in the adverse events for Study 275-08-001. Any event existing prior to the initiation of study treatment that was aggravated after initiation of study treatment was handled as a new event. The investigator assessed the severity of each AE as follows:
  Mild: No disruption of normal daily activities; Moderate: Affected normal daily activities; Severe: Inability to perform daily activities.
  A serious adverse event is an AE that results in death, is life-threatening, requires or prolongs inpatient hospitalization, results in an ongoing or significant incapacity or interferes substantially with normal life functions, or causes a congenital anomaly or birth defect.
Time Frame: From the first dosing of this study up to 12 weeks (84 days) after the last dosing. The dosing was allowed until launch of certolizumab pegol for RA in Japan. The maximum duration on study drug was 204 weeks.
Population: All participants who received at least one study drug administration were included in the safety analysis population (SAF).
Measure: Number; unit: participants
Arm/Group | Discontinued Non-responders 200 mg | Completed Non-responders 200 mg | Completed Responders 200 mg | Completed Responders 400 mg
Number analyzed (Participants) | 81 | 19 | 93 | 92
participants
  Any adverse event | 77 | 18 | 92 | 90
  Mild adverse events | 20 | 4 | 36 | 33
  Moderate adverse events | 47 | 12 | 47 | 45
  Severe adverse events | 10 | 2 | 9 | 12
  Serious adverse events (SAE) | 21 | 4 | 20 | 23
  Serious adverse events leading to death | 1 | 0 | 0 | 0
  Non-fatal serious adverse events | 21 | 4 | 20 | 23
  Adverse events leading to withdrawal | 13 | 2 | 9 | 12
  Infections induced by pathogen in study drug | 0 | 0 | 0 | 0
  Overdoses | 0 | 0 | 0 | 0
  Adverse events occurring within 2 hours of dosing | 1 | 0 | 0 | 0

2. Secondary Outcome: Percentage of Participants With American College of Rheumatology 20% (ACR20) Response
Description: A participant was an ACR20 responder if the following 3 criteria for improvement from Baseline (before study drug administration in Study 275-08-001) were met:
  * ≥ 20% improvement in 68 tender joint count;
  * ≥ 20% improvement in 66 swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of arthritis pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI));
    * C-Reactive Protein (CRP).
Time Frame: Baseline (of Study 275-08-001), Week 24, Week 52 and at the final assessment (maximum was 208 weeks)
Population: The full analysis set (FAS) included all randomized participants who received at least one dose of study drug with at least one post-baseline efficacy data point. Last observation carried forward (LOCF) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Discontinued Non-responders 200 mg | Completed Non-responders 200 mg | Completed Responders 200 mg | Completed Responders 400 mg
Number analyzed (Participants) | 81 | 19 | 93 | 92
percentage of participants
  Week 24 | 71.6 [60.5 to 81.1] | 68.4 [43.4 to 87.4] | 96.8 [90.9 to 99.3] | 98.9 [94.1 to 100.0]
  Week 52 | 76.5 [65.8 to 85.2] | 84.2 [60.4 to 96.6] | 98.9 [94.2 to 100.0] | 94.6 [87.8 to 98.2]
  Final Assessment | 80.2 [69.9 to 88.3] | 89.5 [66.9 to 98.7] | 95.7 [89.4 to 98.8] | 94.6 [87.8 to 98.2]

3. Secondary Outcome: Percentage of Participants With American College of Rheumatology 50% (ACR50) Response
Description: A participant was an ACR50 responder if the following 3 criteria for improvement from Baseline (before study drug administration in Study 275-08-001) were met:
  * ≥ 50% improvement in 68 tender joint count;
  * ≥ 50% improvement in 66 swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of arthritis pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI));
    * C-Reactive Protein (CRP).
Time Frame: Baseline (of Study 275-08-001), Week 24, Week 52 and at the final assessment (maximum was 208 weeks)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Discontinued Non-responders 200 mg | Completed Non-responders 200 mg | Completed Responders 200 mg | Completed Responders 400 mg
Number analyzed (Participants) | 81 | 19 | 93 | 92
percentage of participants
  Week 24 | 42.0 [31.1 to 53.5] | 36.8 [16.3 to 61.6] | 83.9 [74.8 to 90.7] | 82.6 [73.3 to 89.7]
  Week 52 | 48.1 [36.9 to 59.5] | 57.9 [33.5 to 79.7] | 87.1 [78.5 to 93.2] | 88.0 [79.6 to 93.9]
  Final Assessment | 60.5 [49.0 to 71.2] | 57.9 [33.5 to 79.7] | 86.0 [77.3 to 92.3] | 85.9 [77.0 to 92.3]

4. Secondary Outcome: Percentage of Participants With American College of Rheumatology 70% (ACR70) Response
Description: A participant was an ACR70 responder if the following 3 criteria for improvement from Baseline (before study drug administration in Study 275-08-001) were met:
  * ≥ 70% improvement in 68 tender joint count;
  * ≥ 70% improvement in 66 swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of arthritis pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI));
    * C-Reactive Protein (CRP).
Time Frame: Baseline (of Study 275-08-001), Week 24, Week 52 and at the final assessment (maximum was 208 weeks)
Population: The full analysis set (FAS) included all randomized participants who received at least one dose of study drug, with at least one post-baseline efficacy data point. Last observation carried forward (LOCF) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Discontinued Non-responders 200 mg | Completed Non-responders 200 mg | Completed Responders 200 mg | Completed Responders 400 mg
Number analyzed (Participants) | 81 | 19 | 93 | 92
percentage of participants
  Week 24 | 14.8 [7.9 to 24.4] | 26.3 [9.1 to 51.2] | 60.2 [49.5 to 70.2] | 47.8 [37.3 to 58.5]
  Week 52 | 30.9 [21.1 to 42.1] | 31.6 [12.6 to 56.6] | 64.5 [53.9 to 74.2] | 57.6 [46.9 to 67.9]
  Final Assessment | 44.4 [33.4 to 55.9] | 31.6 [12.6 to 56.6] | 65.6 [55.0 to 75.1] | 62.0 [51.2 to 71.9]

5. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS) 28
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables:
  * 28 tender joint count;
  * 28 swollen joint count;
  * Erythrocyte sedimentation rate (ESR);
  * Patient's global assessment of disease activity.
  To obtain the tender joint count and swollen joint count, 28 joints of the shoulder, elbow, wrist, metacarpophalangeal joints, thumb interphalangeal joints, proximal interphalangeal joints, and knee joints were examined.
  The data before study drug administration of 275-08-001 Study was utilized for Baseline.
  DAS28(ESR) scores range from 0 to approximately 10, with the upper bound dependent on the highest possible ESR. A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score of 3.2 or less indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline (of Study 275-08-001), Week 24, Week 52 and at the final assessment (maximum was 208 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Discontinued Non-responders 200 mg | Completed Non-responders 200 mg | Completed Responders 200 mg | Completed Responders 400 mg
Number analyzed (Participants) | 81 | 19 | 93 | 92
units on a scale
  Week 24 | -2.28 (1.27) | -2.32 (1.25) | -3.24 (1.11) | -3.23 (1.24)
  Week 52 | -2.65 (1.44) | -2.34 (0.96) | -3.51 (1.15) | -3.21 (1.29)
  Final Assessment | -2.98 (1.82) | -2.67 (1.44) | -3.49 (1.27) | -3.46 (1.31)

6. Secondary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS)
Description: X-ray images of extremities (posteroanterior views of both hands and dorsoplantar views of both feet) were independently assessed by at least two radiographic readers.
  The degree of joint destruction was graded by assessing bone erosion in 44 joints and joint space narrowing (JSN) in 42 joints.
  The joint erosion score is a summary of erosion severity in 32 joints of the hands and 12 joints in the feet. Each joint was scored, according to the surface area involved, from 0 (no erosion) to 5 (complete collapse of bone). The score for erosion ranges from 0 to 160 in the hands and from 0 to 120 in the feet (the maximum erosion score for a joint in the foot is 10). The JSN score summarizes the severity of JSN in 30 joints of the hands and 12 joints of the feet. JSN, including subluxation, was scored from 0 (normal) to 4 (complete loss of joint space, bony ankylosis, or luxation), with a maximum JSN score of 168. The mTSS ranges from 0 (normal) to 448 (worst).
Time Frame: Baseline (of Study 275-08-001), Week 0 (of this study) and Week 100
Population: Full analysis set with available mTSS data. Linear extrapolation method was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Discontinued Non-responders 200 mg | Completed Non-responders 200 mg | Completed Responders 200 mg | Completed Responders 400 mg
Number analyzed (Participants) | 64 | 16 | 86 | 83
units on a scale
  Change from Baseline to Week 0 | 1.48 (2.70) | 1.69 (2.29) | 0.71 (2.75) | 0.08 (1.83)
  Change from Baseline to Week 100 (N=61, 16, 83, 83 | 5.13 (11.76) | 4.97 (8.79) | 3.77 (12.43) | 2.12 (9.55)

ADVERSE EVENTS:
Time Frame: From the first dosing of this study up to 12 weeks (84 days) after the last dosing. The dosing was allowed until launch of certolizumab pegol for RA in Japan. The maximum duration on study drug was 204 weeks.
Description: All participants who received at least one study drug administration were included in the safety analysis population (SAF).
Arm/Group | Discontinued Non-responders 200 mg | Completed Non-responders 200 mg | Completed Responders 200 mg | Completed Responders 400 mg
Serious Adverse Events (participants affected / at risk) | 21/81 | 4/19 | 20/93 | 23/92
Other Adverse Events (participants affected / at risk) | 77/81 | 18/19 | 91/93 | 90/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Discontinued Non-responders 200 mg (N=81) | Completed Non-responders 200 mg (N=19) | Completed Responders 200 mg (N=93) | Completed Responders 400 mg (N=92)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Pyomyositis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1
Infective tenosynovitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Atypical mycobacterial infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Computerised tomogram thorax abnormal (Investigations) | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 4
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Dementia (Nervous system disorders) | 0 | 0 | 0 | 1
Facial palsy (Nervous system disorders) | 0 | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 2
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Laryngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Abortion induced (Surgical and medical procedures) | 0 | 0 | 1 | 0
Removal of internal fixation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Toe operation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Discontinued Non-responders 200 mg (N=81) | Completed Non-responders 200 mg (N=19) | Completed Responders 200 mg (N=93) | Completed Responders 400 mg (N=92)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 1 | 8 | 5
Vertigo (Ear and labyrinth disorders) | 2 | 2 | 2 | 2
Anovulatory cycle (Endocrine disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 3 | 0 | 5 | 3
Conjunctivitis allergic (Eye disorders) | 8 | 0 | 8 | 8
Diabetic retinopathy (Eye disorders) | 2 | 1 | 0 | 0
Dry eye (Eye disorders) | 2 | 2 | 4 | 2
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1 | 0 | 3
Constipation (Gastrointestinal disorders) | 10 | 2 | 2 | 9
Dental caries (Gastrointestinal disorders) | 8 | 1 | 9 | 6
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 6 | 9
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Duodenal polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 6 | 2
Gastric ulcer (Gastrointestinal disorders) | 2 | 1 | 0 | 2
Gastritis (Gastrointestinal disorders) | 5 | 2 | 3 | 7
Gingivitis (Gastrointestinal disorders) | 0 | 2 | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 1 | 4 | 3
Periodontitis (Gastrointestinal disorders) | 5 | 2 | 8 | 4
Reflux oesophagitis (Gastrointestinal disorders) | 2 | 1 | 3 | 6
Stomach discomfort (Gastrointestinal disorders) | 2 | 0 | 6 | 6
Stomatitis (Gastrointestinal disorders) | 7 | 1 | 3 | 8
Vomiting (Gastrointestinal disorders) | 0 | 3 | 3 | 6
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 3 | 1 | 2 | 2
Cyst (General disorders) | 0 | 1 | 1 | 0
Injection site reaction (General disorders) | 6 | 0 | 1 | 1
Pyrexia (General disorders) | 4 | 1 | 2 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 6 | 1 | 10 | 7
Hepatic steatosis (Hepatobiliary disorders) | 6 | 0 | 5 | 4
Seasonal allergy (Immune system disorders) | 5 | 1 | 10 | 6
Contrast media allergy (Immune system disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 10 | 4 | 14 | 8
Cellulitis (Infections and infestations) | 0 | 1 | 2 | 3
Cystitis (Infections and infestations) | 7 | 2 | 6 | 4
Gastroenteritis (Infections and infestations) | 4 | 1 | 9 | 6
Herpes simplex (Infections and infestations) | 1 | 1 | 1 | 3
Herpes zoster (Infections and infestations) | 2 | 2 | 3 | 4
Influenza (Infections and infestations) | 7 | 1 | 9 | 7
Localised infection (Infections and infestations) | 0 | 1 | 1 | 0
Nasal vestibulitis (Infections and infestations) | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 41 | 12 | 53 | 45
Onychomycosis (Infections and infestations) | 0 | 2 | 3 | 3
Pharyngitis (Infections and infestations) | 15 | 1 | 18 | 10
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 3
Sialoadenitis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 4 | 1 | 2 | 5
Tinea pedis (Infections and infestations) | 5 | 0 | 4 | 9
Upper respiratory tract infection (Infections and infestations) | 15 | 3 | 20 | 20
Urinary tract infection (Infections and infestations) | 3 | 1 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 5 | 2
Oral herpes (Infections and infestations) | 6 | 0 | 7 | 6
Arthropod sting (Injury, poisoning and procedural complications) | 4 | 1 | 3 | 2
Chillblains (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 5 | 2
Contusion (Injury, poisoning and procedural complications) | 9 | 1 | 12 | 6
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 2
Device failure (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1
Bone fissure (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 1
Blood pressure increased (Investigations) | 0 | 1 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 | 0 | 6 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 7 | 8
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 6 | 4 | 10 | 13
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 6 | 3
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 3 | 2 | 5
Sciatica (Nervous system disorders) | 0 | 1 | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 5
Psychosomatic disease (Psychiatric disorders) | 0 | 1 | 0 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 6
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 8 | 7
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 4 | 5
Dermatitis contact (Skin and subcutaneous tissue disorders) | 7 | 0 | 6 | 6
Eczema (Skin and subcutaneous tissue disorders) | 9 | 2 | 14 | 12
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 4 | 4 | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 7 | 1 | 7 | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 5 | 3 | 7 | 8
Asteatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3
Hypertension (Vascular disorders) | 5 | 2 | 9 | 11
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication to seek patent protection.